CLINICAL TRIAL: NCT02293798
Title: Circumferential Periareolar Mastopexy Using SERI Surgical Scaffold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Mofid MD (Individual)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Mark Mofid MD, Principal Investigator, Mofid, Mehrdad Mark, M.D.
Organization: Mofid, Mehrdad Mark, M.D. (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 820
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Mastopexy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SERI (Experimental): Subjects receiving SERI for mastopexy
  Interventions: Device: silk surgical scaffold

INTERVENTIONS:
Device: silk surgical scaffold — surgical implant
  Other Names: SERI surgical scaffold

SUMMARY:
The purpose of this study is to evaluate the clinical performance of SERI® Surgical Scaffold to maintain the size of the areola by providing additional soft tissue support after circumferential periareolar mastopexy.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 years or older desiring a reduction in size of nipple areola complex
* Be in good health and suited to general anesthesia and planned treatments
* Non smokers
* If the subject is of childbearing potential, have a urine pregnancy test evaluated as negative (assessed at baseline examination (Visit 1), agree to use contraception as prevention to avoid pregnancy during the study period
* Previous augmentation with silicone-filled or saline-filled breast implants or patients desiring periareolar mastopexy
* Requiring surgery for ptotic breasts

Exclusion Criteria:

* BMI (Body Mass Index) that is ≥ 30 kg/m2
* Active smoker or have smoked within 6 weeks prior to screening/qualification visit (Visit 1)
* Pregnant or nursing
* Advanced fibrocystic disease considered to be premalignant without accompanying subcutaneous mastectomy
* Previous mastectomy or lumpectomy
* Abscess or infection in the body at the time of enrollment
* Had any disease, including uncontrolled diabetes (e.g., HbAIc > 8%), that is clinically known to impact wound healing ability. For example: collagen-vascular, connective tissue or autoimmune disorders (e.g., Systemic Lupus, Rheumatoid Arthritis, Scleroderma)
* Subjects with diagnosed diabetes must have HbAIc ≤ 8% within 3 months of enrollment
* Is taking medications known to impair wound healing (e.g. corticosteroids, chemotherapeutic agents etc.,)
* Bleeding disorders (e.g., Hemophilia, von Willebrand Disease) including the following medications & supplements: Warfarin, platelet inhibitors (e.g. NSAIDs or Clopidogrel) not stopped within 2 weeks of the operation and herbal supplements known to predispose to bleeding (e.g. Gingko and Ginseng)
* Showed tissue characteristics that were clinically incompatible with mammaplasty, such as tissue damage resulting from radiation, inadequate tissue, compromised vascularity or ulceration
* Had, or was under treatment for, any condition that may have constituted an unwarranted surgical risk (e.g., unstable cardiac or pulmonary problems)
* History of prior implantation of any surgical scaffold (e.g., synthetic mesh, acellular dermal matrix, or biologic mesh) in the breast
* Implantation of any non-SERI® surgical scaffold (e.g., synthetic mesh, acellular dermal matrix, or biologic mesh) during the study period
* Be currently enrolled in another clinical study of an implanted device in the breast or plan to enroll in another clinical study within the study period, which could affect wound healing in the breast repair site and/or would not allow the patient to attend all study visits as outlined within this protocol
* Product contraindications for use of SERI® Surgical Scaffold per the supplied package insert (e.g., hypersensitivity to silk)
* Show psychological characteristics that may have been incompatible with the surgical procedure and the prosthesis, such as inappropriate attitude or motivation (e.g., body dysmorphic disorder)
* Active alcohol/substance abuse problem or have had a relapse within 1 year prior to screening/qualification visit (Visit 1)
* Was not willing to undergo further surgery for revision, if medically required

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: SERI Mesh
Period: Overall Study
Arm/Group | SERI
Started | 13; 26 SERI Mesh (2 units of SERI Mesh placed in each patient)
Completed | 13; 26 SERI Mesh (2 units of SERI Mesh placed in each patient)
Not Completed | 0; 0 SERI Mesh

BASELINE CHARACTERISTICS:
Arm/Group | SERI
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 32.85 [24 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Areolar Dilation of up to 6mm at 12 Months
Description: areolar dilation of up to 6mm
Time Frame: 12 months after SERI implantation
Measure: Count of Participants; unit: Participants
Arm/Group | SERI
Number analyzed (Participants) | 13
Participants | 13

ADVERSE EVENTS:
Arm/Group | SERI
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No